CLINICAL TRIAL: NCT07285538
Title: A Prospective Interventional Study of Stereotactic Body RadioTherapy (SBRT) With Continuous Tracking for Inoperable Patients With Primary and Secondary Renal Cancer (SBRTRC)
Brief Title: Stereotactic Body RadioTherapy With Continuous Tracking for Primary and Secondary Renal Cancer
Acronym: SBRTRC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Nadia Di Muzio, Professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRTRC
Record Dates: First submitted 2025-11-26; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Renal Cancer; Renal Secondary Cancer; Stereotactic Body Radiotherapy
Keywords: Renal primary tumors; Renal secondary tumors; stereotactic body radiotherapy; stereotactic ablative radiotherapy; Renal toxicity
MeSH Terms: conditions — Kidney Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: A total of 60 patients are expected to be enrolled in this prospective, non-randomized study. For the sample size calculation, a power of 80% and a significance level (α) of 5% are set. The hypothesis is that the proportion of patients free from ≥G2 toxicity 3 years after the end of treatment is less than or equal to 13% which is inferior to the ≥G2 toxicity of 36% registered in the FASTRACK II trial. Considering a simple proportion study a total of 60 patients are required, including an additional 20% to compensate for potential drop-outs (relative to toxicity outcome). In case of reaching toxicity and local control objectives the study will be closed after another two years of follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective, interventional, monocentric, clinical study of SBRT for primary/secondary renal tumor (Experimental): SBRT to renal lesions will be delivered using 1-5 fractions. Dose and fractionation options will attempt to keep the biologically effective dose (BED) to ≥80 Gy assuming an α/β ratio of 10 due to association with improved local control. Established dosing regimens include:
  * 25-26 Gy in 1 fraction, for lesion in the greatest diameter (or sum of diameters in case of multiple lesions) up to 4 cm of maximum diameter
  * 42-48 Gy in 3-4 fractions, for lesion in the greatest diameter (or sum of diameters in case of multiple lesions) up to 6 cm of maximum diameter
  * 40-50 Gy in 5 fractions, for lesion larger than 6 cm in the greatest diameter (or sum of diameters in case of multiple lesions) For multi-fraction dosing, treatment will be delivered on consecutive or alternate days.
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — SBRT for primary or secondary renal tumors, delivering from 25-26 Gy/1 fraction to 42-48 Gy/3-4 fractions or 40-50 Gy/5 fractions (according to tumor size), using CyberKnife

SUMMARY:
This is a prospective, interventional, monocentric, clinical study of Stereotactic Body Radiation Therapy (SBRT) for primary or secondary renal tumors, delivering from 25-26 Gy/1 fraction to 42-48 Gy/3-4 fractions or 40-50 Gy/5 fractions (standard prescriptions for the internationl guidelines, according to tumor size), using a robotic accelerator -CyberKnife® (Accuray, Sunnyvale, CA)-, with fiducial-tracking, to observe the acute and late toxicity reduction (as primary objectives), due to the maximum precision of the treatment. Secondary objectives are Local Relpase-Free Survival (LRFS), Regional Relapse-Free Survival (RRFS), Distant Metastasis-Free Survival (DMFS), Disease-Free Survival (DFS), Cancer Specific Survival (CSS), Overall Survival (OS) and Quality-of-Life (QoL). A total of 60 participants are expected to be enrolled over four years, and the follow-up of enrolled patients will be three years.

DETAILED DESCRIPTION:
Renal Cell Carcinoma (RCC) is the eighth most common cancer diagnosed in Europe, with a rising incidence, particularly in old patients. The standard of care for operable patients with primary RCC is surgical resection, however, not all patients are suitable candidates for surgery. Alternative approaches, such as thermal ablation, present significant limitations, as reduced efficacy for lager tumors (>3-4 cm) and those located near the renal hilum.

Traditionally, Radiotherapy (RT) has not been considered an effective treatment for RCC due to its perceived radioresistance. High dose radiation therapy RCC leads to both direct cancer cell death and indirect cancer death from vasculature disruption.

The paradigm of radioresistance has shifted significantly with the advent of stereotactic body radiotherapy/ ablative radiotherapy (SBRT/SABR), which has demonstrated promising efficacy in local control while preserving renal function. The radiosensitivity varies in laboratory studies, with low α/β values (2.6 Gy - 6.9 Gy), thus RCC's lines are more responsive to increased radiation fraction size.

SBRT is non-invasive, delivers high doses with precision, using a steep dose gradient over a small number of treatment sessions. This approach has recently demonstrated promising local control (LC), and acceptable toxicity, even for large tumors.

IROCK (the International Radiosurgery Consortium of the Kidney) included 223 patients pooled from nine institutions, with a median follow up of 30 months. No difference in LC and toxicity was observed between patients receiving single fraction SBRT at 25 Gy (range 14-26 Gy) and multiple fractions SBRT at a median of 40 Gy (range 24-70 Gy) in four fractions was observed.

In 2022, IROCK reported the 5-year outcomes of 190 patients with primary RCC. The 7-year cumulative local failure rate was 8.4%, with no significant difference in the incidence of grade ≥2 between single fraction SBRT (5%) and multi-fraction SBRT (6%).

The TransTasman Radiation Oncology Group (TROG) 15.03 FASTRACK II trial was a non-randomized, phase 2, multicenter study with 71 pts enrolled, and 70 underwent SBRT. Treatment was delivered according to tumor size, with 23 patients (33%) received a single- fraction dose of 26 Gy (for tumors ≤ 4 cm) and 47 patients received 42 Gy in 3 fractions (for tumors >4 and ≤10 cm). Median follow up was 43 months. Local Control was 100%, with no observed local failures during the study protocol. Cancer specific survival was 100%, while freedom from distant failure was 97% at 36 months. Overall Survival was 82% at 36 months. SBRT was well tolerated with no grade 4 or 5 adverse events. The systematic review conducted for the International Society of Stereotactic Radiosurgery (ISRS) guidelines analyzed 36 studies with 822 patients. The median LC was 94.1 % (range 70-100%), 5-year progression-free survival was 80.5 % (range 72-92%), and 5- year Overall Survival was 77.2 %. SBRT was associated with minimal impact on renal function, with only a 3.9% of patients requiring post treatment dialysis across studies. Abancourt et al. analyzed 144 patients treated between 2008 and 2020, mainly with 26 Gy/ 1 fraction and 42 Gy/ 3 fractions, and with a 43 month median follow-up (IQR 24-81.2) local control at 5 years was 96%. Overall survival was 58 months and 5-year cumulative incidence of cancer related deaths was 8% (95% CI 3-15%). As much as 49% of patients experienced at least one toxicity, of which 32% were grade 1, 14% grade 2 and 1% grade 3. Two patients (1%) underwent dialysis. Median eGFR loss was 7 ml/min (IQR -17; 0) at the last follow-up.

The proposed clinical study involves a cutting-edge dose delivery method and a precise treatment planning. The high-dose conformation and real-time imaging accuracy for target identification and adjustment during treatment ensure the validity of this approach.

The treatment will be performed according to current guidelines. For primary disease definitive radiation therapy using SBRT will be considered as a treatment option for non-optimal surgical candidates, for patients with T1 tumors (<10 cm in diameter, according to FASTRACK II trial). SBRT will be delivered using 1-5 fractions. Dose and fractionation options will attempt to keep the biologically effective dose (BED) to ≥80 Gy assuming an α/β ratio of 10 due to association with improved local control.

This is a prospective, interventional, monocentric, clinical study of SBRT for primary or secondary renal tumors, delivering from 25-26 Gy/1 fraction to 40-50 Gy/5 fractions (according to tumor size), using CyberKnife with fiducial-tracking. The primary objective is acute and late toxicity reduction, due to the maximum precision of the treatment. Secondary objectives concern loco-regional and distant control, overall and specific survival, quality-of-life.

The study plans to enroll a total of 60 patients, needed for the ≥ G2 toxicity analysis , according to the study design, and with 20% compensation for potential drop-outs.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or clinical diagnosis of primary or secondary kidney tumors
2. Patients aged ≥18 years
3. Signed informed consent
4. Tumor up to 10 cm in the greatest diameter (sum of diameters in case of multiple lesions)
5. PS (ECOG) ≤2
6. No prior local radiotherapy
7. Fertile women using contraception methods previously initiated (a pregnancy test will be prescribed)

Exclusion Criteria:

1. Patients aged < 18 years
2. Tumors > 10 cm
3. PS ECOG ≥3
4. Psychiatric or other disorders that may prevent the patient from signing informed consent
5. Previous invasive cancer, except for skin cancer (excluding melanoma) unless the patient has been disease-free for at least 3 years (e.g., carcinoma in situ of the oral cavity or bladder)
6. Pregnant women
7. Collagen diseases
8. Sjogren's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2033-01-15 (Estimated); Study Completion 2033-01-15 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 3 months
  Acute toxicity grade ≥2 as the maximum toxicity value at 3 months after the completion of radiotherapy treatment evaluated with Common Toxicity Criteria For Adverse Events (CTCAE) scale, v6.0, with 5 grades, from 0 = no change, to 5 = death for toxicity
Late toxicity | 3 years
  Late toxicity grade ≥2 as the maximum toxicity value at 3 years after the completion of radiotherapy treatment evaluated with Common Toxicity Criteria For Adverse Events (CTCAE) scale, v6.0, with 5 grades, from 0 = no change, to 5 = death for toxicity

SECONDARY OUTCOMES:
Local control of the treated lesion (LC) | 3 years
  Local control of the treated site expressed in terms of local recurrence rate
Local Relapse-Free Survival (time to local recurrence, LRFS) | 3 years
  From the date of radiotherapy end until the date of local relapse, assessed up to 3 years
Regional Relapse-Free Survival (RRFS) | 3 years
  From the date of radiotherapy end until the date of regional relapse, assessed up to 3 years
Distant Metastases-Free Survival (DMFS) | 3 years
  From the date of radiotherapy end until the date of distant metasis diagnosis, assessed up to 3 years
Disease-Free Survival (local, regional, distant, DFS) | 3 years
  From the date of radiotherapy end until the date of first, any ( local, regional, distant) relapse, assessed up to 3 years
Cancer Specific Survival (CSS) | 3 years
  From the date of radiotherapy end until the date of death from renal cancer, assessed up to 3 years
Overall Survival (OS) | 3 years
  From the date of radiotherapy end until the date of death from any cause, assessed up to 3 years

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed with tumor specific quality of life questionnaires | 3 years
  Quality of life (QoL) related to treatment using the European Organisation for Research and Treatment of Cancer (EORTC) Italian version of quality-of-life core QLQ-C30 questionnaire completed before treatment, at the end of treatment, and at 1, 3, 6, 12, 18, 24, 36 months after SBRT.
Organ motion | Perioperative/periprocedural
  Modeling of organ movement during treatment
Clinical and dosimetric prognostic factors | 3 years
  Identification of clinical, imaging, and laboratory prognostic factors for an aggressive phenotype of kidney cancer and for toxicity.
Radiomics | 3 years
  Evaluation of radiomic characteristics: Mathematical extraction of the spatial distribution of signal intensities and pixel interrelationships of medical images of the patients, to quantify textural information resampled according to International Biomarker Standardization Initiative (IBSI).

CONTACTS AND LOCATIONS:
Overall Officials: Nadia G Di Muzio, Prof., Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- Department of Radiation Oncology, IRCCS San Raffaele Scientific Institute, Milan, Milano (MI), Italy

REFERENCES:
- [Result] Abancourt L, Ali M, Quivrin M, Wallet J, Schick U, Ingrosso G, Supiot S, Franzese C, Scorsetti M, Kerkmeijer L, Fodor A, Muzio ND, Jousset N, Boisserie T, Detti B, Nicosia L, Alongi F, Trippa F, Leleu T, Dessoude L, Terlizzi M, Blanchard P, Scher N, Toledano A, Baude J, Lartigau E, Barthoulot M, Siva S, Pasquier D. Results of Stereotactic Body Radiation Therapy for Primary Renal Cell Carcinoma in a Large Multicenter Series. Eur Urol Oncol. 2025 Jun;8(3):774-781. doi: 10.1016/j.euo.2025.01.001. Epub 2025 Feb 7. PMID 39920013
- [Result] Siva S, Bressel M, Sidhom M, Sridharan S, Vanneste BGL, Davey R, Montgomery R, Ruben J, Foroudi F, Higgs B, Lin C, Raman A, Hardcastle N, Hofman MS, De Abreu Lourenco R, Shaw M, Mancuso P, Moon D, Wong LM, Lawrentschuk N, Wood S, Brook NR, Kron T, Martin J, Pryor D; FASTRACK II Investigator Group. Stereotactic ablative body radiotherapy for primary kidney cancer (TROG 15.03 FASTRACK II): a non-randomised phase 2 trial. Lancet Oncol. 2024 Mar;25(3):308-316. doi: 10.1016/S1470-2045(24)00020-2. PMID 38423047
- [Result] Siva S, Ali M, Correa RJM, Muacevic A, Ponsky L, Ellis RJ, Lo SS, Onishi H, Swaminath A, McLaughlin M, Morgan SC, Cury FL, Teh BS, Mahadevan A, Kaplan ID, Chu W, Grubb W, Hannan R, Staehler M, Warner A, Louie AV. 5-year outcomes after stereotactic ablative body radiotherapy for primary renal cell carcinoma: an individual patient data meta-analysis from IROCK (the International Radiosurgery Consortium of the Kidney). Lancet Oncol. 2022 Dec;23(12):1508-1516. doi: 10.1016/S1470-2045(22)00656-8. Epub 2022 Nov 16. PMID 36400098
- [Result] Siva S, Louie AV, Warner A, Muacevic A, Gandhidasan S, Ponsky L, Ellis R, Kaplan I, Mahadevan A, Chu W, Swaminath A, Onishi H, Teh B, Correa RJ, Lo SS, Staehler M. Pooled analysis of stereotactic ablative radiotherapy for primary renal cell carcinoma: A report from the International Radiosurgery Oncology Consortium for Kidney (IROCK). Cancer. 2018 Mar 1;124(5):934-942. doi: 10.1002/cncr.31156. Epub 2017 Dec 20. PMID 29266183
- [Result] Ali M, Mooi J, Lawrentschuk N, McKay RR, Hannan R, Lo SS, Hall WA, Siva S. The Role of Stereotactic Ablative Body Radiotherapy in Renal Cell Carcinoma. Eur Urol. 2022 Dec;82(6):613-622. doi: 10.1016/j.eururo.2022.06.017. Epub 2022 Jul 14. PMID 35843777
- [Result] Siva S, Chesson B, Bressel M, Pryor D, Higgs B, Reynolds HM, Hardcastle N, Montgomery R, Vanneste B, Khoo V, Ruben J, Lau E, Hofman MS, De Abreu Lourenco R, Sridharan S, Brook NR, Martin J, Lawrentschuk N, Kron T, Foroudi F. TROG 15.03 phase II clinical trial of Focal Ablative STereotactic Radiosurgery for Cancers of the Kidney - FASTRACK II. BMC Cancer. 2018 Oct 23;18(1):1030. doi: 10.1186/s12885-018-4916-2. PMID 30352550
- [Result] Rich BJ, Noy MA, Dal Pra A. Stereotactic Body Radiotherapy for Localized Kidney Cancer. Curr Urol Rep. 2022 Dec;23(12):371-381. doi: 10.1007/s11934-022-01125-6. Epub 2022 Nov 16. PMID 36383304
- [Result] Moreno-Olmedo E, Sabharwal A, Das P, Dallas N, Ford D, Perna C, Camilleri P. The Landscape of Stereotactic Ablative Radiotherapy (SABR) for Renal Cell Cancer (RCC). Cancers (Basel). 2024 Jul 27;16(15):2678. doi: 10.3390/cancers16152678. PMID 39123406
- [Result] Siva S, Louie AV, Kotecha R, Barber MN, Ali M, Zhang Z, Guckenberger M, Kim MS, Scorsetti M, Tree AC, Slotman BJ, Sahgal A, Lo SS. Stereotactic body radiotherapy for primary renal cell carcinoma: a systematic review and practice guideline from the International Society of Stereotactic Radiosurgery (ISRS). Lancet Oncol. 2024 Jan;25(1):e18-e28. doi: 10.1016/S1470-2045(23)00513-2. PMID 38181809
- [Result] Palumbo C, Pecoraro A, Knipper S, Rosiello G, Luzzago S, Deuker M, Tian Z, Shariat SF, Simeone C, Briganti A, Saad F, Berruti A, Antonelli A, Karakiewicz PI. Contemporary Age-adjusted Incidence and Mortality Rates of Renal Cell Carcinoma: Analysis According to Gender, Race, Stage, Grade, and Histology. Eur Urol Focus. 2021 May;7(3):644-652. doi: 10.1016/j.euf.2020.05.003. Epub 2020 May 23. PMID 32456993
- [Result] Capitanio U, Bensalah K, Bex A, Boorjian SA, Bray F, Coleman J, Gore JL, Sun M, Wood C, Russo P. Epidemiology of Renal Cell Carcinoma. Eur Urol. 2019 Jan;75(1):74-84. doi: 10.1016/j.eururo.2018.08.036. Epub 2018 Sep 19. PMID 30243799